CLINICAL TRIAL: NCT00143988
Title: Heart Rate and Blood Pressure Response During Exercise and Sexual Activity in Normotensive and Hypertensive Volunteers
Acronym: SEXERRCISE
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sebastian T. Palmeri, MD - Principal Investigator, UMDNJ-Robert Wood Johnson Medical School
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 3255; investigator initiated trial
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-08

CONDITIONS: Heart Rate; Blood Pressure
Keywords: Blood Pressure; Heart Rate; Sexual Activity
MeSH Terms: conditions — Sexual Behavior | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Treadmill Test exertion females
  Interventions: Behavioral: Treadmill testing
- Treadmill test exertion males
  Interventions: Behavioral: Treadmill testing
- Sexual activity exertion females
  Interventions: Behavioral: Ambulatory Blood Pressure and Heart Rate Monitoring
- Sexual activity exertion males
  Interventions: Behavioral: Ambulatory Blood Pressure and Heart Rate Monitoring

INTERVENTIONS:
Behavioral: Treadmill testing — Patients will have a exercise stress test using a Bruce protocol during which time heart rates and blood pressures will be monitored and the patient's percieved exertion level monitored and recorded
  Other Names: Quinton treadmill will be used
  Groups: Treadmill Test exertion females; Treadmill test exertion males
Behavioral: Ambulatory Blood Pressure and Heart Rate Monitoring — Patients will wear an ambulatory blood pressure monitor and an heart rate monitor during one sexual encounter.
  Other Names: Space Labs ambulatory BP monitor; Polar heart rate monitor
  Groups: Sexual activity exertion females; Sexual activity exertion males

SUMMARY:
The purpose of this study is to determine the amount of cardiac work as measured by heart rate and blood pressure during physical exertion compared to sexual activity.

DETAILED DESCRIPTION:
Physical exertion will be measured by a standardized treadmill test. Sexual activity will be performed in the study subject's home with his/her spouse or regular partner. Each study subject will wear a blood pressure and heart rate monitor at home during their sexual activity and will be asked to complete a one page diary upon completion of the activity. Normotensive and subject with mild hypertension will be studied to determine if hypertensive subjects have a relatively greater increase in their blood pressure during either physical exercise or sexual activity.

ELIGIBILITY:
Inclusion Criteri

1) Male or female age 40-80

Exclusion Criteria

1. Current sexual partner less than six months duration or sexually inactive patients defined as engaging in sexual intercourse less than one time monthly
2. Uncontrolled hypertension (resting blood pressure >160/100); secondary hypertension; renal failure (serum creatinine >3.0); congestive heart failure (NYHA functional Class III-IV); acute coronary syndrome; PCI or open heart surgery within past 3 months; cerebrovascular disease within the past 6 months and any other major medical or psychiatric disorder.

   * Individuals who regularly (more than 3 times weekly) perform rigorous physical exercise.
   * Individuals unable to perform an exercise treadmill stress test.
   * Lack of informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women over the age of 40 who are sexually active
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2004-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
physical stress during exercise | during one measured encounter

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Palmeri, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Mittleman MA, Maclure M, Tofler GH, Sherwood JB, Goldberg RJ, Muller JE. Triggering of acute myocardial infarction by heavy physical exertion. Protection against triggering by regular exertion. Determinants of Myocardial Infarction Onset Study Investigators. N Engl J Med. 1993 Dec 2;329(23):1677-83. doi: 10.1056/NEJM199312023292301. PMID 8232456
- [Background] Tofler GH, Stone PH, Maclure M, Edelman E, Davis VG, Robertson T, Antman EM, Muller JE. Analysis of possible triggers of acute myocardial infarction (the MILIS study). Am J Cardiol. 1990 Jul 1;66(1):22-7. doi: 10.1016/0002-9149(90)90729-k. PMID 2193495
- [Background] Muller JE, Mittleman MA, Maclure M, Sherwood JB, Tofler GH. Triggering myocardial infarction by sexual activity. Low absolute risk and prevention by regular physical exertion. Determinants of Myocardial Infarction Onset Study Investigators. JAMA. 1996 May 8;275(18):1405-9. doi: 10.1001/jama.275.18.1405. PMID 8618365
- [Background] Hellerstein HK, Friedman EH. Sexual activity and the postcoronary patient. Arch Intern Med. 1970 Jun;125(6):987-99. No abstract available. PMID 4951941
- [Background] Bohlen JG, Held JP, Sanderson MO, Patterson RP. Heart rate, rate-pressure product, and oxygen uptake during four sexual activities. Arch Intern Med. 1984 Sep;144(9):1745-8. PMID 6476990
- [Background] Green AW. Sexual activity and the postmyocardial infarction patient. Am Heart J. 1975 Feb;89(2):246-52. doi: 10.1016/0002-8703(75)90055-1. No abstract available. PMID 805515
- [Background] Nemec ED, Mansfield L, Kennedy JW. Heart rate and blood pressure responses during sexual activity in normal males. Am Heart J. 1976 Sep;92(3):274-7. doi: 10.1016/s0002-8703(76)80106-8. PMID 949020
- [Background] Mann S, Craig MW, Gould BA, Melville DI, Raftery EB. Coital blood pressure in hypertensives. Cephalgia, syncope, and the effects of beta-blockade. Br Heart J. 1982 Jan;47(1):84-9. doi: 10.1136/hrt.47.1.84. PMID 6119996
- [Background] Drory Y, Shapira I, Fisman EZ, Pines A. Myocardial ischemia during sexual activity in patients with coronary artery disease. Am J Cardiol. 1995 Apr 15;75(12):835-7. doi: 10.1016/s0002-9149(99)80425-1. No abstract available. PMID 7717293
- [Background] Standards for adult exercise testing laboratories. American Heart Association Subcommittee on Rehabilitation, Target Activity Group. Circulation. 1979 Feb;59(2):421A-430A passim. No abstract available. PMID 759014